CLINICAL TRIAL: NCT01889212
Title: Imaging With 11C-erlotinib PET/CT to Identify Responders to Erlotinib Treatment in NSCLC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to technical problems
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1-10-72-19-12
Record Dates: First submitted 2013-06-03; First posted 2013-06-28 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2013-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NSCLC, erlotinib treatment, 11C-erlotinib PET/CT (Experimental)
  Interventions: Other: 11C-erlotinib PET/CT

INTERVENTIONS:
Other: 11C-erlotinib PET/CT

SUMMARY:
New treatment strategies have been developed in lung cancer targeting the Epidermal Growth Factor Receptor (EGFR). Patients with an activating mutation in the EGFR have high responds rates to the treatment and should be treated with a EGFR inhibitor as first line of treatment. Some wild type patients do as well respond but selection of these patients is more difficult.

Erlotinib has been labeling with 11C and used as a new PET tracer. Accumulation of the tracer (11C-erlotinib) in tumors has showed promising results for selection of responders.

The investigators now want to conduct a larger clinical study to evaluate if accumulation of tracer on a pre-treatment 11C-erlotinib PET/CT can predict responds to erlotinib.

ELIGIBILITY:
Inclusion Criteria:

* Lung Cancer patients with non-small cell histology and stage IV disease who are candidate for erlotinib treatment as first/ second/ third line of treatment

Exclusion Criteria:

* pregnancy
* severe dyspnoea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Accumulation of 11c-erlotinib in tumors before and after treatment with erlotinib | From date of inclusion until the date of first documented progression on the erlotinib treatment or date of death, whichever came first, assessed up to 30 months
  Accumulation of 11c-erlotinib in tumors will be correlated to PFS on erlotinib treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Meldgaard, Ph.D MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Deparment of oncology, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/22095231